CLINICAL TRIAL: NCT07051694
Title: Exploratory Study on Transcutaneous Auricular Vagus Nerve Stimulation as Adjuvant Treatment for Sepsis Patients
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation as Adjuvant Treatment for Sepsis Patients
Acronym: TaVNS-Sepsis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Tan Liang, Clinical Professor, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIIT2024050
Record Dates: First submitted 2025-06-03; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Sepsis
Keywords: sepsis; transcutaneous auricular vagus nerve stimulation
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS group (Experimental): transcutaneous auricular vagus nerve stimulation twice a day for 7 consecutive days.
  Interventions: Device: taVNS
- sham-taVNS group (Sham Comparator): sham transcutaneous auricular vagus nerve stimulation twice a day for 7 consecutive days.
  Interventions: Device: sham-taVNS

INTERVENTIONS:
Device: taVNS — Transcutaneous Auricular Vagus Nerve Stimulation
  Arms: taVNS group
Device: sham-taVNS — sham transcutaneous auricular vagus nerve stimulation
  Arms: sham-taVNS group

SUMMARY:
The goals of this randomized clinical trial are to investigate the effects of transcutaneous auricular vagus nerve stimulation (taVNS) combined with standard intensive care on systemic organ function in septic patients, and exploring its potential mechanisms for improving overall outcomes in sepsis.The main question it aims to answer is whether taVNS can reduce the severity of sepsis patients by ameliorating systemic inflammation.Participants will receive standard intensive care treatment and be randomized to receive the taVNS or sham taVNS as adjuvant treatment twice a day for 7 consecutive days. Several evaluations will be done before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Sepsis was diagnosed per the Sepsis-3 criteria (SCCM/ESICM 2016) as infection with SOFA score ≥ 2
* ICU admission within 7 days after sepsis onset
* Informed consent was obtained from patients/guardians

Exclusion Criteria:

* severe ARDS defined by PaO₂/FiO₂ ≤100 mmHg with PEEP ≥5 cm H₂O
* HR>120 per minute
* epinephrine or norepinephrine >1ug/kg/min
* severe underlying pulmonary diseases including interstitial lung disease, -
* diffuse alveolar hemorrhage, severe asthma, or lung cancer
* taVNS contraindications: existing pacemakers, cochlear implants, or other active implantable electronic medical devices
* dermatologic or infectious disorders affecting the auricular region
* pregnancy or lactation
* participation in other clinical trials
* inability to remain motionless during treatment (e.g., due to epilepsy or Parkinson's disease)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
SOFA socre | Baseline and Day 8
  The total SOFA score is obtained by adding the scores of the six systems: respiratory, coagulation, liver, cardiovascular, central nervous, and renal. The SOFA score ranges from 0 to 24, with a higher score indicating more severe organ dysfunction.

SECONDARY OUTCOMES:
blood | Baseline and Day 8
  Routine complete blood count
Glasgow coma scale | Baseline and Day 8
  pecific scoring criteria were established for eye opening, verbal response, and motor response, with maximum scores of 4, 5, and 6 points respectively. A higher score indicating better condition.
tidal volume | Baseline and Day 8
  tested by mechanical ventilation
vasoactive-intropic score | Baseline and Day 8
  VIS can intuitively reflect the degree of dependence of sepsis patients on vasoactive drugs, providing a quantitative indicator for clinicians. It helps to more accurately assess the condition of sepsis, evaluate the therapeutic effect and predict the prognosis. The larger the value, the more severe the condition.
Arterial blood gas (ABG) analysis | Baseline and Day 8
  Arterial blood gas (ABG) analysis
fraction of inspiration O2 | Baseline and Day 8
  tested by mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Army Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
ResMan, http://www.medresman.org.cn/login.aspx
Supporting Information: ICF
Time Frame: 1year after publishing this research paper
Access Criteria: anyone who are intrested in this research
URL: http://www.medresman.org.cn/login.aspx

DOCUMENTS (1):
  • Informed Consent Form (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT07051694/ICF_000.pdf